CLINICAL TRIAL: NCT04547725
Title: Complete Cytoreductive Surgery With Combined Intraperitoneal and Systemic Chemotherapies for Gastric Adenocarcinoma Patients With Limited Peritoneal Carcinomatosis: an Open-label Two-stage Phase II Trial
Brief Title: Complete Cytoreduction Followed by IP and Systemic Chemotherapies for Gastric Cancer With Peritoneal Carcinomatosis
Acronym: CRS-IP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202006125RINC
Record Dates: First submitted 2020-09-02; First posted 2020-09-14 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Gastric Cancer; Peritoneal Carcinomatosis
Keywords: gastric cancer; peritoneal carcinomatosis; cytoreductive surgery; intraperitoneal chemotherapy
MeSH Terms: conditions — Stomach Neoplasms; Peritoneal Neoplasms

STUDY DESIGN:
Intervention Model Description: Complete cytoreductive surgery followed by intraperitoneal and systemic chemotherapies
Masking Description: Arm-A: resectable advanced gastric adenocarcinoma with limited PC (PCI ≤ 10) Arm-B: resectable advanced gastric adenocarcinoma with positive peritoneal wash cytology (CY1/P0)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CRS-IP (Arm-A) (Experimental): Stage IV gastric cancer with limited peritoneal carcinomatosis (peritoneal carcinomatosis index [PCI] ≤ 10)
  Interventions: Other: CRS followed by IP and systemic chemotherapies
- CRS-IP (Arm-B) (Experimental): Stage IV gastric cancer with positive peritoneal wash cytology (CY1/P0)
  Interventions: Other: CRS followed by IP and systemic chemotherapies

INTERVENTIONS:
Other: CRS followed by IP and systemic chemotherapies — Complete cytoreductive surgery (CRS) + normothermic intraperitoneal chemotherapy (N-IPEC) + systemic chemotherapy

SUMMARY:
Background: Approximately 15% of gastric adenocarcinoma patients presents with peritoneal carcinomatosis (PC) at the first encounter and is regarded as an unresectable and end-stage disease. The recommended treatment with palliative chemotherapy alone yields a poor clinical efficacy. Emerging evidences suggest the survival benefits of complete cytoreductive surgery (CRS) combined with normothermic intraperitoneal chemotherapy (N-IPEC) for gastric adenocarcinoma with limited PC.

Objective: To evaluate the 6-month disease control rate (DCR) of complete CRS combined with N-IPEC and systemic chemotherapy for gastric adenocarcinoma with limited PC.

Patients and methods: Patients having gastric adenocarcinoma with PCI ≤ 10 (Arm-A) or positive peritoneal wash cytology (CY1/P0) (Arm-B) will be enrolled. Patients with other distant metastasis, including brain, lung, liver, bone, will be excluded. All patients should undergo ≥ D2 gastrectomy and complete CRS followed by N-IPEC (paclitaxel] and systemic chemotherapy (high-dose fluorouracil and cisplatin [P-HDFL], or capecitabine and oxaliplatin [CAPOX]). N-IPEC (paclitaxel) will be administered in combination with systemic P-HDFL or CAPOX on day 1,8,15 or day 1,8 for each cycle, respectively. The disease status will be evaluated every 12 weeks based on the computed tomography scan, and the clinical evaluation (outpatient follow-up) will be performed every 2 weeks for whom receiving P-HDFL and every 3 weeks for whom receiving CAPOX. Patients will receive maximal 6 cycles N-IPEC with P-HDFL or 8 cycles N-IPEC with CAPOX. After N-IPEC is discontinued, P-HDFL or CAPOX will be continued alone until disease progression or death. The primary endpoint of this study is 6-month DCR, and the secondary endpoints include 6-month response rate for ascites, 1-year progression-free survival (PFS) and overall survival (OS), 3-year PFS and OS, and safety profiles. Based on Simon's minimax two-stage design, this trial will be carried out in two stages. In stage I, a total number of 13 (Arm-A) / 16 (Arm-B) patients is accrued. If there are ≤ 6 (Arm-A) / ≤ 14 (Arm-B) progression-free among these 13 (Arm-A) / 16 (Arm-B) patients, the study will be early stopped. Otherwise, additional 17 (Arm-A) / 2 (Arm-B) patients will be accrued in stage II, resulting in a total number sample size of 30 (Arm-A) / 18 (Arm-B).

Expected result: A ≥ 75% (Arm-A) / ≥ 95% (Arm-B) 6-month DCR could be achieved for gastric adenocarcinoma patients with limited PC (Arm-A) / with CY1P0 (Arm-B) via this treatment strategy (complete CRS + N-IPEC + P-HDFL or CAPOX) -i.e., if there are ≥ 21 (Arm-A) / ≥ 16 (Arm-B) progression-free among the 30 (Arm-A) / 18 (Arm-B) enrolled patients, we will reject the null hypothesis and claim that the treatment is promising.

DETAILED DESCRIPTION:
Background: Approximately 15% of gastric adenocarcinoma patients presents with peritoneal carcinomatosis (PC) at the first encounter and is regarded as an unresectable and end-stage disease. The recommended treatment with palliative chemotherapy alone yields a poor clinical efficacy and long-term prognosis. Emerging evidences suggest the survival benefits of complete cytoreductive surgery (CRS) combined with intraperitoneal chemotherapy (IP) for gastric adenocarcinoma with limited PC. Previous studies focused on the CRS combined with hyperthermic IP chemotherapy (HIPEC); however, the high morbidity and mortality rates of HIPEC have raised a safety concern and limited the clinical application. The normothermic IP chemotherapy (N-IPEC), on the other hand, is a safer and gentler type of IP chemotherapy, and has gained in popularity and been evaluated in many recent clinical trials. The criteria for patient selection and standard protocol of complete CRS combined with N-IPEC and systemic chemotherapy remain to be determined. Moreover, treatment efficacy regarding this strategy is still suboptimal.

Objective: To evaluate the 6-month disease control rate (DCR) of complete CRS combined with N-IPEC (paclitaxel) and systemic chemotherapy (high-dose fluorouracil and cisplatin; [P-HDFL], or capecitabine and oxaliplatin [CAPOX]) for gastric adenocarcinoma patients with limited PC (peritoneal carcinomatosis index [PCI] ≤ 10) (Arm-A) or positive peritoneal wash cytology (CY1/P0) (Arm-B).

Patients and methods: Patients having resectable advanced gastric adenocarcinoma with limited PC (PCI ≤ 10) (Arm-A) or positive peritoneal wash cytology (CY1/P0) (Arm-B) will be enrolled. Patients with distant metastasis other than PC, including brain, lung, liver, bone, will be excluded. All patients should undergo D2 or more extensive gastrectomy and complete CRS followed by N-IPEC (paclitaxel) and systemic chemotherapy (P-HDFL or CAPOX). N-IPEC with paclitaxel 20 mg/m2 will be administered in combination with systemic P-HDFL or CAPOX on day 1,8,15 or day 1,8 for each cycle, respectively. Peritoneal cytology will be collected at the surgery and on day 1 of each treatment cycle. The disease status and ascites amount will be evaluated every 12 weeks based on the computed tomography scan, and the clinical evaluation (outpatient follow-up) will be performed every 2 weeks for whom receiving P-HDFL and every 3 weeks for whom receiving CAPOX. Patients will receive maximal 6 cycles N-IPEC with P-HDFL (total 18 courses of N-IPEC) or 8 cycles N-IPEC with CAPOX (total 16 courses of N-IPEC). After N-IPEC is discontinued, P-HDFL or CAPOX will be continued alone until disease progression or death. The primary endpoint of this study is 6-month DCR, and the secondary endpoints include 6-month response rate for ascites, 1-year progression-free survival (PFS) and overall survival (OS), 3-year PFS and OS, and safety profiles. Based on Simon's minimax two-stage design, this trial will be carried out in two stages. In stage I, a total number of 13 (Arm-A) / 16 (Arm-B) patients is accrued. If there are ≤ 6 (Arm-A) / ≤ 14 (Arm-B) progression-free among these 13 (Arm-A) / 16 (Arm-B) patients, the study will be early stopped. Otherwise, additional 17 (Arm-A) / 2 (Arm-B) patients will be accrued in stage II, resulting in a total number sample size of 30 (Arm-A) / 18 (Arm-B).

Expected result: A ≥ 75% (Arm-A) / ≥ 95% (Arm-B) 6-month DCR could be achieved for gastric adenocarcinoma patients with limited PC (Arm-A) / with CY1P0 (Arm-B) via this treatment strategy (complete CRS + N-IPEC + P-HDFL or CAPOX) -i.e., if there are ≥ 21 (Arm-A) / ≥ 16 (Arm-B) progression-free among the 30 (Arm-A) / 18 (Arm-B) enrolled patients, we will reject the null hypothesis and claim that the treatment is promising.

ELIGIBILITY:
[Inclusion criteria]

1. Age 20 to 75 years old.
2. Blood tests:

   1. White blood cells > 4,000/mm3, neutrophils > 1,500/mm3, platelets > 100,000/mm3.
   2. Serum creatinine < 1.5 mg/dl or creatinine clearance > 60 ml/min.
   3. Serum bilirubin < 2 mg/dl.
3. Eastern Cooperative Oncology Group (ECOG) Performance Status = 0 or 1.
4. Not legal incapacity.
5. Newly diagnosed gastric adenocarcinoma, including Siewert III adenocarcinoma of the cardia, with limited peritoneal carcinomatosis (PCI ≤ 10) or positive peritoneal wash cytology (CY1/P0) .

[Exclusion criteria]

1. Prior malignancy within 3 years or with detectable signs of recurrence.
2. Newly diagnosed gastric adenocarcinoma having been treated by preoperative systemic or intraperitoneal chemotherapy.
3. Presence of comorbidities, including liver cirrhosis (≥ Child B), decompensated heart failure (New York Heart Association [NYHA] Class III or IV congestive heart failure), poorly-controlled chronic obstructive pulmonary disease.
4. ≥ American Society of Anesthesiologists Classification (ASA Class) Class 3.
5. Pregnancy or breastfeeding.
6. Intolerability of chemotherapeutic agents in this study:

   1. N-IPEC paclitaxel (all patients).
   2. Capecitabine or oxaliplatin (patients who receive CAPOX regimen).
   3. Cisplatin or 5-fluorouracil (patients who receive P-HDFL regimen).
7. Distant metastases (e.g. liver, lung, bone) except for the peritoneum, intra-abdominal lymph node, and ovary.
8. Extensive PC (PCI > 10).
9. Siewert I or II adenocarcinoma of the cardia.
10. Other patients inappropriate for this study in the opinion of the investigators.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2020-09-16 (Actual); Primary Completion 2026-03-16 (Estimated); Study Completion 2028-09-16 (Estimated)

PRIMARY OUTCOMES:
6-month disease control rate | 6 months
  The 6-month disease control rate is defined as the percentage of patients with no occurrence of radiological PD (per RECIST 1.1), clinical PD (based on investigator's judgement), or death from any cause, after 24 weeks (~ 6 months) from the beginning of combined IP and systemic chemotherapies.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | 3 years
  The 1-year and 3-year PFS, defined as the time from the date of enrollment until the date of PD or death from any cause, whichever is earliest, during the first and the first three years of the study, respectively.
Overall survival (OS) | 3 years
  The 1-year and 3-year OS, defined as the time from the date of enrollment until the date of death from any cause, during the first and the first three years of the study, respectively.
6-month response rate for ascites. | 6 months
  The 6-month response rate for ascites: the percentage of patients with complete disappearance (CR-ascites) or a dramatic decrease in ascites (PR-ascites) at the time when the 6-month disease control rate is evaluated.
Safety evaluation | 9 months
  Safety endpoints, including surgery-related complications, toxicities of chemotherapy, and intraperitoneal port/catheter-related complications, will be evaluated throughout the treatment period (at every follow-up visit), and then 30 days and 90 days after the treatment period is discontinued.

CONTACTS AND LOCATIONS:
Overall Officials: I-Rue Lai, MDPHD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No